CLINICAL TRIAL: NCT04355533
Title: Seroprevalence and Antibody Profiling Against SARS-CoV2 in Children and Their Parents
Brief Title: Immunity Against SARS-CoV2 in Children and Their Parents / COVID-19
Acronym: PED-COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Commissariat A L'energie Atomique (Other Government); Institut Pasteur (Industry); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP200467; 2020-A00999-30 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: COVID-19 Infection
Keywords: Child; COVID-19 infection; immune response; healthy carrier
MeSH Terms: conditions — COVID-19 | interventions — Serologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Hospitalized children or consulting at hospital (Experimental)
  Interventions: Biological: serology test; Biological: nasopharyngeal swab; Biological: rectal swab; Biological: saliva sample
- Parents of one included child (Experimental)
  Interventions: Biological: serology test; Biological: nasopharyngeal swab; Biological: saliva sample
- Children with potential COVID disease during the first wave (Experimental)
  Interventions: Biological: serology test; Biological: nasopharyngeal swab; Biological: rectal swab; Biological: saliva sample
- Children SARS-coV2 positive (Experimental)
  Interventions: Biological: serology test; Biological: nasopharyngeal swab; Biological: rectal swab; Biological: saliva sample
- Person living under the same roof as children included in the study (Experimental)
  Interventions: Biological: serology test; Biological: nasopharyngeal swab; Biological: rectal swab; Biological: saliva sample

INTERVENTIONS:
Biological: serology test — volume according to child weight
Biological: nasopharyngeal swab — nasopharyngeal swab for PCR
Biological: rectal swab — rectal swab for PCR
  Arms: Children SARS-coV2 positive; Children with potential COVID disease during the first wave; Hospitalized children or consulting at hospital; Person living under the same roof as children included in the study
Biological: saliva sample — for biocollection

SUMMARY:
The purpose of this study is to provide data on the proportion of seroconverted children and their immune status. It will also provide insight into the number of children currently infected at each time point including healthy carriers. Investigators will provide similar data on their parents in an ancillary study.

DETAILED DESCRIPTION:
The fraction of undiagnosed but likely to transmit the virus is a critical epidemiological characteristic that modulates the epidemic potential of SARS-CoV2. To adapt the epidemy control, it is essential to study the immunoprotection of the general population. A crucial question is the study of pauci or asymptomatic subjects, and in particular children who make mild forms, because they could act as a real reservoir for the spread of the virus. The serological study is essential in this context.

The serologic test Abbott will be used to study immunoprevalence. Institut Pasteur has validated test using neutralizing Ab. CEA will used a antibodies and antigen test.

ELIGIBILITY:
Inclusion Criteria:

For hospitalized children or consulting at hospital

* any child over 7 days old and under 17 years old in consultation or hospitalized for at most 4 days at AP-HP or CH Cayenne; Or any child over 7 days old and under 17 years old with a positive PCR at home, with an attending physician in a participating centre
* Parent's agreement for blood, saliva and stool samples
* Optional parent's agreement for nasopharynx swab
* Optional parent's agreement for follow-up if PCR+
* With an Health insurance

For children with potential COVID disease during the first wave

* Any child over 7 days old and under 17 years, seropositive during the first wave
* Or any child over 7 days old and under 17 years, with a previous inflammatory clinical disease potentially linked to SARS-cov2
* With an Health insurance

Parent of the enrolled child

* One parent of the enrolled child on ped-covid
* Agreement for blood and saliva samples
* Optional agreement for nasopharynx swab
* Optional parent's agreement for follow-up if PCR+
* With an Health insurance

For children SARS-coV2 positive

* any child less then 18 years old
* infected by SARS-coV2
* Parent's agreement for blood, saliva samples
* Optional parent's agreement for nasopharynx swab
* With health insurance

For people living under the same roof of a child included in the study

* any child or adult living under the same roof of a child SARS-coV2 positive and included in the study
* With health insurance

Exclusion Criteria:

For hospitalized children or consulting at hospital

* child younger than 7 days
* Refusal of parent
* Refusal of child
* No health insurance

Min Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1056 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
Seroconversion against SARS-CoV2 in children | at inclusion
  serology

SECONDARY OUTCOMES:
Measure of Ab antiN and Ab anti-S1/2 | at inclusion
  Serology in children
Neutralization activity | at inclusion
  Serology in children
Positive qPCR in children | at inclusion
  in children, qualitative and quantitative measure , in nasopharynx, saliva and stool
correlation between different Ab and qPCR and neutralization activity | at inclusion
  in children, qualitative and quantitative measure , in nasopharynx, saliva and stool, Ab anti-N, Ab anti-S1/2, neutralization serum
Protective immunity | Day 3
  Serology, measure of Ab in PCR positive children
Protective immunity | Day 7
  Serology, measure of Ab in PCR positive children
Protective immunity | Day 15
  Serology, measure of Ab in PCR positive children
Protective immunity | Day 45
  Serology, measure of Ab in PCR positive children
Protective immunity | At 6 months
  Serology, measure of Ab in PCR positive children
Protective immunity | At 12 months
  Serology, measure of Ab in PCR positive children
Duration of viral carriage in stool, saliva and or nasopharynx | until 45 days if persistence of positive qPCR
  Sars-Cov2 PCR in PCR positive children
Correlation between antibody profile and viral clearance | until 45 days post onset
  Serology in PCR positive children
Ab profile and memory of immunity | At Day 3
  Immune cells in positive PCR children
Ab profile and memory of immunity | At Day 7
  Immune cells in positive PCR children
Ab profile and memory of immunity | At Day 15
  Immune cells in positive PCR children
Ab profile and memory of immunity | At Day 45
  Immune cells in positive PCR children
Ab profile and memory of immunity | At 6 months
  Immune cells in positive PCR children
Ab profile and memory of immunity | At 12 months
  Immune cells in positive PCR children
saliva biofluid characteristics of COVID-19 infected | Until 1 year follow-up
  viral content (qPCR and immunodetection); presence of IgG, M, and A
Presence of the virus | Until 1 year follow-up
  In PCR positive children: nasopharynx, saliva, stool
Reinfection | Until 1 year follow-up
  In PCR positive children: occurrence of reinfection, immunity responses during reinfection and potential mutations of the virus
Transmission of the virus to the family | until 45 days follow-up
  symptomatic, virological and serological follow-up
Immune response | At inclusion
  In children COVID+ during the first wave :immune response few months after the infection
Mucosal immunity | Until 1 year follow-up
  In PCR positive children: Ab anti-SARS-cov2 in nasopharynx samples
seroconversion against SARS-CoV2 in parents | at inclusion
  Ancillary study: Serology in parents
Measure of Ab antiN and Ab anti-S1 and neutralization activity | at inclusion
  Ancillary study: Serology in parents
Positive qPCR in parents | at inclusion
  Ancillary study: in parents, qualitative and quantitative measure , in nasopharynx, saliva
Correlation between different Ab and qPCR | at inclusion
  Ancillary study: in parents, qualitative and quantitative measure , in nasopharynx, saliva, Ab anti-N, Ab anti-S1, neutralization serum
Correlation between antibody profile and viral clearance | until 45 days post onset
  Ancillary study: Serology in PCR positive parents
Ab profile and memory of immunity | at Day 3
  Ancillary study: Immune cells in positive PCR parents
Ab profile and memory of immunity | at Day 7
  Ancillary study: Immune cells in positive PCR parents
Ab profile and memory of immunity | at Day 15
  Ancillary study: Immune cells in positive PCR parents
Ab profile and memory of immunity | at Day 45
  Ancillary study: Immune cells in positive PCR parents
Ab profile and memory of immunity | at 6 months
  Ancillary study: Immune cells in positive PCR parents
Ab profile and memory of immunity | at 12 months
  Ancillary study: Immune cells in positive PCR parents
Saliva biofluid characteristics of COVID-19 infected | Until 1 year follow-up
  in positive PCR parents: viral content (qPCR and immunodetection); presence of IgG, M, and A
Presence of the virus | Until 45 days follow-up
  in positive PCR parents: nasopharynx, saliva
Mucosal immunity | Until 1 year follow-up
  in positive PCR parents: Ab anti-SARS-cov2 in nasopharynx samples
Reinfection | Until 1 year follow-up
  in positive PCR parents: occurrence of reinfection, immunity responses during reinfection and potential mutations of the virus

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle SERMET-GAUDELUS, MD, PhD, Principal Investigator — Assistance Publique-Hôpitaux de Pars
Locations (1):
- Hôpital necker Enfants-Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Delaunay-Moisan A, Guilleminot T, Semeraro M, Briand N, Bader-Meunier B, Berthaud R, Morelle G, Quartier P, Galeotti C, Basmaci R, Benoist G, Gajdos V, Lorrot M, Rifai M, Crespin M, M'Sakni Z, Padavia F, Savetier-Leroy C, Lorenzi M, Maurin C, Behillil S, de Pontual L, Elenga N, Bouazza N, Moltrecht B, van der Werf S, Leruez-Ville M, Sermet-Gaudelus I. Saliva for molecular detection of SARS-CoV-2 in pre-school and school-age children. Environ Microbiol. 2022 Oct;24(10):4725-4737. doi: 10.1111/1462-2920.16151. Epub 2022 Aug 12. PMID 36065993